CLINICAL TRIAL: NCT03722342
Title: A Phase 1b, Open-Label, Safety and Tolerability Study of TTAC-0001 in Combination With Pembrolizumab in Patients With Recurrent Glioblastoma
Brief Title: TTAC-0001 and Pembrolizumab Combination phase1b Trial in Recurrent Glioblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PharmAbcine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PMC_TTAC-0001_04
Record Dates: First submitted 2018-07-03; First posted 2018-10-26 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — olinvacimab

STUDY DESIGN:
Intervention Model Description: This was mTPI design to start with optimal dose and next dose level is selected accroding to DLT occurrance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TTAC-0001 and pembrolizumab (Experimental): TTAC-0001 and pembrolizumab combination therapy will be administered.
  Interventions: Drug: TTAC-0001 and pembrolizumab combination

INTERVENTIONS:
Drug: TTAC-0001 and pembrolizumab combination — * Investigational product (IP): TTAC-0001 and Pembrolizumab (Merck, Keytruda®)
  * Treatment groups: 3 dose levels
    * Dose level 1 (optimal starting dose): TTAC-0001 12 mg/kg on D1, D8 and D15 + Pembrolizumab 200 mg on D1
    * Dose level 2 (first escalation dose): TTAC-0001 16 mg/kg on D1, D8 and D15 + Pembrolizumab 200 mg on D1
    * Dose level 0 (de-escalation dose): TTAC-0001 8 mg/kg on D1, D8 and D15 + Pembrolizumab 200 mg on D1
  * Cycle: 3 weeks (21 days per cycle)

SUMMARY:
This is a phase 1b, open-Label clinical trial to determine the safety and tolerability and to establish a preliminary recommended Phase 2 dose (RP2D) of TTAC-0001 administered in combination with pembrolizumab in patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with primary glioblastoma by histopathological examination and confirmed recurrent glioblastoma by magnetic resonance imaging (MRI) scans after completing standard of care (Stupp protocol) concomitant temozolomide chemotherapy with radiotherapy (CCRT)
2. At least one confirmed measurable lesion by RANO criteria
3. Karnofsky Performance Status (KPS) ≥80
4. A person who satisfies the following criteria in haematologic, renal, and hepatic function tests performed within 7 days prior to screening:

   1. Haematologic tests

      * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
      * Platelets ≥ 100 x 109/L
      * Haemoglobin ≥ 9.0 g/dL
   2. Blood coagulation tests

      * Prothrombin time (PT) ≤ 1.5 x Upper limit of normal (ULN)
      * Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
   3. Hepatic function tests

      * Total bilirubin ≤ 1.5 x UNL
      * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastasis)
   4. Renal function test

      * ≤1.5 × ULN or creatinine clearance (CrCl) ≥30 mL/min for patient with creatinine levels >1.5 × institutional ULN
5. At least 12 weeks of expected survival time
6. The patient (or legally acceptable representative if applicable) is able and willing to provide written informed consent for the trial

Exclusion Criteria:

1. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. (Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ [e.g., breast carcinoma, cervical cancer in situ] controlled by curative therapy are not excluded)
2. Has received prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
3. Has a history of (non-infectious) pneumonitis/interstitial lung diseases that required steroids or current pneumonitis/interstitial lung disease
4. Has an active infection requiring systemic therapy
5. Uncontrolled hypertension (systolic blood pressure [SBP]> 150 or diastolic blood pressure [DBP]> 90 mmHg)
6. Uncontrolled seizures
7. Class III or IV heart failure by New York Heart Association (NYHA) classification
8. Has oxygen-dependent chronic disease
9. Active psychiatric disorder (schizophrenia, major depressive disorder, bipolar disorder etc.). Treated depression with ongoing antidepressant medication is not an exclusion
10. History of abdominal fistula or gastrointestinal perforation within 6 months prior to start of study drug
11. History of serious gastrointestinal haemorrhage within 6 months prior to start of study drug
12. History of severe arterial thromboembolic event within 12 months of start of study drug
13. Serious grade 4 venous thromboembolic event including pulmonary embolism
14. History of hypertensive crisis or hypertensive encephalopathy
15. History of posterior reversible encephalopathy syndrome
16. Planned surgery within 4 weeks post last dose
17. Moderate to severe proteinuria as demonstrated by urine dipstick for proteinuria ≥2+. For patients with ≥2+ proteinuria on dipstick urinalysis, a urine protein: creatinine (UPC) ratio will be determined, or a 24-hour urine collection will be done. Patients with a UPC ratio <1 or a 24-hour urine protein <1 gram are eligible
18. Requiring therapeutic anticoagulation with warfarin at baseline; patients must be off warfarin or warfarin-derivative anticoagulants for at least 7 days prior to starting study drug; however, therapeutic or prophylactic therapy with low-molecular weight heparin is allowed
19. Not recovered below National Cancer Institute-Common Terminology for Adverse Events (NCI-CTCAE) grade 1 or baseline from AEs due to previous therapy (patient with ≤ Grade 2 neuropathy or alopecia may be eligible)
20. Treatment with systemic chemotherapy, hormonal therapy, immunotherapy or biologic therapy within 2 weeks prior to the baseline visit
21. Undergone major surgery requiring general anaesthesia or a respiratory assistance device within 4 weeks prior to the baseline visit (within 2 weeks for video-assisted thoracoscopic surgery [VATS] or open-and-closed [ONC] surgery)
22. Treated with other investigational drugs within 4 weeks prior to the baseline visit for this study
23. Pregnant* or lactating females, and females/males of childbearing potential who do not agree to a reliable and adequate method of contraception
24. A known history of severe drug hypersensitivity or hypersensitivity to a therapy similar to the study drugs
25. Unable to participate in the trial according to the investigator's decision
26. Previous therapy with vascular endothelial growth factor (VEGF)-targeted agents including (but not limited to) bevacizumab
27. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher irAE
28. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
29. Known human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority
30. Known active hepatitis B or hepatitis C infection. No testing for hepatitis B and hepatitis C is required unless mandated by local health authority
31. Have received a live vaccine within 30 days prior to enrollment. Seasonal flu vaccines that do not contain live virus are permitted
32. Have had a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities | During the first cycle (every cycle is 21 days) of treatment
  The frequency and percentage of DLT will be presented by dose level
Adverse events | From the screening visit to the end of treatment visit (time of progressive disease or 2 years)
  The frequency and percentage of AEs will be presented by dose level
Immunogenicity | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Presence anti-drug antibody (ADA) will be listed

SECONDARY OUTCOMES:
Overall response rate | At every 2nd cycles until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years (every cycle is 21 days)
  complete response (CR) or partial response (PR) by RANO criteria
Disease control rate | At every 2nd cycles until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years (every cycle is 21 days)
  complete response (CR), partial response (PR) or stable disease (SD) by RANO criteria
Progression free survival | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Period from the date of the drug administration to the disease progression time point
Overall survival | From screening visit to date of patient's death (assessed up to 2 year after end of treatment visit)
  Period from the date of the drug administration to the patient's death

OTHER OUTCOMES:
Pharmacokinetic parameters - Cmax | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Maximum concentration of drug by dose level
Pharmacokinetic parameters - Cmin | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Minimum concentration of drug by dose level
Pharmacokinetic parameters - AUC0-t | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Area under the curve from baseline to each timepoint by dose level
Pharmacokinetic parameters - Tmax | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Time of Cmax by dose level
Pharmacokinetic parameters - CL | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Clearance by dose level
Pharmacokinetic parameters - Vd | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Volume of distribution by dose level
Pharmacokinetic parameters - Ke | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Elimination rate constant by dose level
Pharmacokinetic parameters - T½ | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Half-life by dose level
Change in concentration of serum angiogenic factor or receptor | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  VEGF, placental growth factor [PLGF], soluble vascular endothelial growth factor receptor [sVEGFR]-2, sVEGFR-1, etc.
DCE-MRI | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  Blood flow parameter - iAUC, K-trans
PD-L1, VEGFR-2 expression level | From screening visit to end of treatment visit (time of progressive disease or 2 years)
  PD-L1, VEGFR-2 expression level in tumour environment such as tumour, tumour vessel and parenchymal tissue

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Austin Hospital, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia